CLINICAL TRIAL: NCT03958877
Title: An Open-Label, Randomized, Multicenter, Active-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, and Efficacy of BIIB017 in Pediatric Subjects Aged 10 to Less Than 18 Years for the Treatment of Relapsing-Remitting Multiple Sclerosis, With Optional Open-Label Extension
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of BIIB017 (Peginterferon Beta-1a) in Pediatric Participants for the Treatment of Relapsing-Remitting Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105MS306; 2018-003008-38 (EudraCT Number); 2023-505624-56 (Other: EU CTIS)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — peginterferon beta-1a; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB017 (peginterferon beta-1a) (Experimental): Participants will receive subcutaneous (SC) injection of BIIB017 (peginterferon beta-1a) 63 microgram (μg) on Day 1, followed by 94 μg at Week 2, followed by 125 μg at Week 4, and then 125 μg SC injection every 2 weeks up to Week 96 in Part 1 of the study. Eligible participants who enter optional Part 2 of the study will receive 125 μg SC injections of BIIB017 every 2 weeks for 96 Weeks.
  Interventions: Drug: BIIB017 (peginterferon beta-1a)
- Avonex (Active Comparator): Participants will receive Avonex (interferon beta type 1a) starting at a dose of 7.5 μg on Day 1, followed by an increase of 7.5 μg each week for 3 weeks, followed by 30 μg intramuscular (IM) injections every week up to Week 96 in Part 1 of the study. Eligible participants who enter optional Part 2 of the study will receive 125 μg SC injections of BIIB017 every 2 weeks for 96 Weeks.
  Interventions: Drug: Interferon beta type 1a

INTERVENTIONS:
Drug: BIIB017 (peginterferon beta-1a) — Administered as specified in the treatment arm
  Other Names: PLEGRIDY
  Arms: BIIB017 (peginterferon beta-1a)
Drug: Interferon beta type 1a — Administered as specified in the treatment arm
  Other Names: Avonex
  Arms: Avonex

SUMMARY:
This study will evaluate the safety, tolerability, and descriptive efficacy of BIIB017 in pediatric participants with relapsing-remitting multiple sclerosis (RRMS) and to assess the pharmacokinetics (PK) of BIIB017 in pediatric participants with RRMS in Part 1. In Part 2, the study will evaluate the long-term safety of BIIB017 and further describe safety and the long-term multiple sclerosis (MS) outcomes after BIIB017 treatment in participants who completed the study treatment at Week 96 in Part 1 of the study.

ELIGIBILITY:
Key Inclusion Criteria:

Part 1:

* Must have a diagnosis of RRMS as defined by the revised consensus definition for pediatric MS.
* Must have an EDSS score between 0.0 and 5.5.
* Must have experienced >= 1 relapse in the 12 months prior to randomization (Day 1) or >= 2 relapses in the 24 months prior to randomization (Day 1) or have evidence of asymptomatic disease activity (Gd-enhancing lesions) on brain MRI in the 6 months prior to randomization (Day 1).

Part 2:

• Participants who completed the study treatment in Part 1 (Week 96 Visit), as per protocol.

Key Exclusion Criteria:

Part 1:

* Primary progressive, secondary progressive, or progressive relapsing MS. These conditions require the presence of continuous clinical disease worsening over a period of at least 3 months. Participants with these conditions may also have superimposed relapses but are distinguished from relapsing participants by the lack of clinically stable periods or clinical improvement.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* Known allergy to any component of Avonex or BIIB017 formulation.
* Occurrence of an MS relapse that has occurred within 30 days prior to randomization (Day 1) and/or the participant has not stabilized from a previous relapse prior to randomization (Day 1).
* Any previous treatment with PEGylated human IFN β-1a.

Part 2:

* Any significant changes in medical history occurring after enrollment in Part 1, including laboratory test abnormalities or current clinically significant conditions that, in the opinion of the Investigator, would have excluded the participant's participation in Part 1. The Investigator must re-assess the participant's medical fitness for participation and consider any factors that would preclude treatment.
* The participant could not tolerate BIIB017 in Part 1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Part 1: Annualized Relapse Rate (ARR) at Week 48 | Week 48
  A multiple sclerosis (MS) relapse is defined as the onset of new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings. ARR is calculated as the total number of relapses in each treatment group adjusted for the duration of study treatment in person-years.
Part 2: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading to Study Treatment Discontinuation | From Week 96 to Week 196
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, or is a medically important event.

SECONDARY OUTCOMES:
Part 1: ARR at Week 96 | Week 96
  An MS relapse is defined as the onset of new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings. ARR is calculated as the total number of relapses in each treatment group adjusted for the duration of study treatment in person-years.
Part 1: Percentage of Participants Free of New or Newly Enlarging T2 Hyperintense Lesions on Brain Magnetic Resonance Imaging (MRI) Scans at Weeks 24, 48, and 96 | Weeks 24, 48, and 96
Part 1: Percentage of Participants Free of New MRI Activity in the Brain (Free of Gadolinium [Gd]-Enhancing Lesions and New or Newly Enlarging T2 Hyperintense Lesions) at Weeks 24, 48, and 96 | Weeks 24, 48, and 96
Part 1: Number of New or Newly Enlarging T2 Hyperintense Lesions on Brain MRI Scans at Weeks 24, 48, and 96 | Weeks 24, 48, and 96
Part 1: Number of Gd-Enhancing Lesions on Brain MRI Scans at Weeks 24, 48, and 96 | Weeks 24, 48, and 96
Part 1: Time to First Relapse | Up to Week 96
Part 1: Percentage of Participants Free of Relapse at Weeks 48 and 96 | Weeks 48 and 96
Part 1: Change from Baseline in Cognition at Weeks 24, 48, 72, and 96 as Measured by the Symbol Digit Modality Test (SDMT) | Baseline, Weeks 24, 48, 72, and 96
  The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0 (worst) to 110 (best) in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution. Higher scores indicate better performance.
Part 1: Change from Baseline in the Expanded Disability Status Scale (EDSS) Score at Weeks 48 and 96 | Baseline, Weeks 48, and 96
  EDSS is based on a standardized neurological exam and focuses on symptoms that commonly occur in MS. Scores range from 0.0 (normal) to 10.0 (death due to MS).
Part 1: Change from Baseline in the Quality of Life as Measured by the Pediatric Quality of Life Inventory (PedsQL) at Weeks 24, 48, 72 and 96 | Baseline, Weeks 24, 48, 72 and 96
  The PedsQL consists of 23 items in four generic score scales: physical functioning, emotional functioning, social functioning, and school functioning that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
Part 1: Area Under the Plasma Concentration-Time Curve from Time Zero to End of Dosing Interval (AUCtau) for BIIB017 | Within 8 hours postdose on Day 1 of Week 1; Within 8 hours, 48 and 120 hours postdose on Day 1 of Week 4; Within 8 hours postdose on Day 1 of Week 24
Part 1: Maximum Observed Plasma Concentration (Cmax) at Steady State for BIIB017 | Within 8 hours postdose on Day 1 of Week 1; Within 8 hours, 48 and 120 hours postdose on Day 1 of Week 4; Within 8 hours postdose on Day 1 of Week 24
Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) at Steady State for BIIB017 | Within 8 hours postdose on Day 1 of Week 1; Within 8 hours, 48 and 120 hours postdose on Day 1 of Week 4; Within 8 hours postdose on Day 1 of Week 24
Part 1: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Study Treatment Discontinuation | Up to Week 100
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, or is a medically important event.
Part 1: Change from Baseline in Height at Weeks 24, 48, 72, 96, and 100 | Baseline, Weeks 24, 48, 72, 96, and 100
Part 1: Change from Baseline in Weight at Weeks 24, 48, 72, 96, and 100 | Baseline, Weeks 24, 48, 72, 96, and 100
Part 1: Change from Baseline in Tanner Score at Weeks 24, 48, 72, 96, and 100 | Baseline, Weeks 24, 48, 72, 96, and 100
  Assessment of Tanner stages (a scale of physical development) will be performed by a medical doctor experienced with this assessment. Tanner score ranges from Stage 1 (childhood) to Stage 5 (full physical maturity). Information regarding Tanner staging will be collected for all male participants with bone age less than (<) 16 years and for female participants who are pre-menarche and have a bone age < 16 years and will be stopped once the participant's bone age reaches greater than or equal to (>=) 16 years or (once the participant is post-menarche. Tanner Score can be omitted if required by country-specific regulations and/or local ethics committees.
Part 1: Number of Participants With Binding and Neutralizing Antibodies to Interferon Beta Type 1a (IFN β-1a) [All Participants] | Up to Week 96
  Presence of IFN β-1a antibodies in human serum will be determined using enzyme-linked immunosorbent assay (ELISA) followed by further characterization and titration of positive samples in a cell-based neutralizing antibody assay.
Part 1: Number of Participants With Binding Antibodies to Peginterferon (PEG) [BIIB017-Treated Participants] | Up to Week 96
  Anti-PEG binding antibodies in human serum will be determined using an ELISA.
Part 1: Change from Baseline in Depression as Assessed by Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) at Weeks 12, 24, 36, 48, 60, 72, 84, 96, and 100 | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, and 100
  MINI-KID is a short (approximately 15 minute) structured diagnostic interview used to assess the presence of 20 diagnostic and statistical manual of mental disorders, 4th Edition (DSM-IV) child and adolescent psychiatric disorders as well as the risk of suicide. The MINI-Kid frames questions in language that is easy for children and adolescents. It consists of 137 questions across 24 modules.
Part 1: Change from Baseline in Blood Pressure at Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100 | Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100
Part 1: Change from Baseline in Pulse Rate at Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100 | Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100
Part 1: Change from Baseline in Body Temperature at Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100 | Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100
Part 1: Change from Baseline in Respiratory Rate at Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100 | Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100
Part 1: Change from Baseline in 12-Lead Electrocardiogram (ECG) Parameters at Weeks 48, 96, and 100 | Baseline (Before dosing), Weeks 48, 96, and 100
Part 1: Percentage of Participants with Changes Over Time in Clinical Laboratory Values | Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and 100
  Clinical laboratory tests include: hematology, chemistry (including liver, renal and thyroid function), and coagulation tests.
Part 2: ARR at Weeks 144 and 192 | Weeks 144 and 192
  An MS relapse is defined as the onset of new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings. ARR is calculated as the total number of relapses in each treatment group adjusted for the duration of study treatment in person-years.
Part 2: Change from Baseline in EDSS Score at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
  EDSS is based on a standardized neurological exam and focuses on symptoms that commonly occur in MS. Scores range from 0.0 (normal) to 10.0 (death due to MS).
Part 2: Change from Baseline in Height at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
Part 2: Change from Baseline in Weight at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
Part 2: Change from Baseline in Tanner Score at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
  Assessment of Tanner stages (a scale of physical development) will be performed by a medical doctor experienced with this assessment. Tanner score ranges from Stage 1 (childhood) to Stage 5 (full physical maturity). Information regarding Tanner staging will be collected for all male participants with bone age < 16 years and for female participants who are pre-menarche and have a bone age <16 years and will be stopped once the participant's bone age reaches >= 16 years or (once the participant is post-menarche. Tanner Score can be omitted if required by country-specific regulations and/or local ethics committees.
Part 2: Number of Participants With Binding and Neutralizing Antibodies to IFN β-1a (All Participants) | Up to Week 192
  Presence of IFN β-1a antibodies in human serum will be determined using ELISA followed by further characterization and titration of positive samples in a cell-based neutralizing antibody assay.
Part 2: Number of Participants With Binding Antibodies to PEG (BIIB017-Treated Participants) | Up to Week 192
  Anti-PEG binding antibodies in human serum will be determined using an ELISA.
Part 2: Change from Baseline in Blood Pressure at Weeks 120,144,168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
Part 2: Change from Baseline in Pulse Rate at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
Part 2: Change from Baseline in Body Temperature at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
Part 2: Change from Baseline in Respiratory Rate at Weeks 120, 144, 168, 192, and 196 | Baseline (Week 96), Weeks 120, 144, 168, 192, and 196
Part 2: Change from Baseline in 12-Lead ECG Parameters at Weeks 144, 192, and 196 | Baseline (Week 96), Weeks 144, 192, and 196
Part 2: Change from Baseline in Depression as Assessed by Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) at Weeks 108, 120, 132, 144,156, 168, 180, 192, and 196 | Baseline (Week 96), Weeks 108, 120, 132, 144,156, 168, 180, 192, and 196
  MINI-KID is a structured diagnostic interview instrument for psychiatric evaluation and outcome tracking. All questions are answered Yes or No.
Part 2: Percentage of Participants with Changes Over Time in Clinical Laboratory Values | Baseline (Week 96), Weeks 108, 120, 132, 144, 156, 168, 180, 192, and 196
  Clinical laboratory tests include: hematology, chemistry (including liver, renal and thyroid function), and coagulation tests.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (65):
- United States (3):
  - UC San Diego Health, La Jolla, California
  - UNC Hospitals, Chapel Hill, North Carolina
  - Meridian Clinical Research, Norfolk, Virginia
- Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires, Buenos Aires, Argentina
- Royal Children's Hospital, Parkville, Victoria, Australia
- Belgium (2):
  - Universitair Ziekenhuis Ghent, Ghent, East Flanders
  - Clinique CHC MontLégia, Liège, Wallonia
- MHATNP 'Sv.Naum', EAD, Sofia, Bulgaria
- Croatia (4):
  - University Hospital Centre Split, Split, Dalmatia
  - Children's Hospital Zagreb, Zagreb
  - Clinical Hospital Center 'Sestre Milosrdnice', Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Fakultni nemocnice Hradec Kralove, Hradec Králové, Czechia
- France (5):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Hopital Purpan, Toulouse, Haute Garonne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
- Germany (4):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - St. Josef-Hospital Universitaetsklinikum, Bochum, North Rhine-Westphalia
  - Charité - Campus Virchow-Klinikum, Berlin
- Greece (2):
  - General Hospital of Larissa, Larissa, Thessaly
  - General Hospital of Thessaloniki 'Hippokration', Thessaloniki
- Hungary (3):
  - Pecsi Tudomanyegyetem KK, Pécs, Baranya
  - Debreceni Egyetem, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem, Budapest
- Israel (2):
  - Hadassah University Hospital - Ein Kerem, Jerusalem, Levant
  - Schneider Children's Medical Center, Petach-Tikva, Tel Aviv
- Italy (3):
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - Azienda Ospedaliera Universitaria 'Federico II', Napoli
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
- Ibn Sina Hospital, Ash Shuwaykh, Shuwaikh, Kuwait
- Portugal (5):
  - Centro Hospitalar e Universitário Lisboa Norte E.P.E., Lisbon, Lisbon District
  - Hospital Beatriz Ângelo, Loures, Lisbon District
  - Hospital de Braga, Braga, Minho
  - Centro Hospitalar e Universitário de Coimbra E.P.E. - Hospital Pediátrico, Coimbra
  - Centro Hospitalar do Porto, E.P.E. - Hospital de Santo António, Porto
- Russia (10):
  - SBEI HPE 'Bashkir State Medical University' of the MoH of the RF, Ufa, Bashkortostan Republic
  - FSBI "Federal Siberian Scientific-Clinical Center of FMBA", Krasnoyarsk, Krasnoyarsk Krai
  - Nebbiolo LLC, Tomsk, Oblast
  - LLC National center for socially significan disease, Saint Petersburg, Sankt-Peterburg
  - SAIH 'Kemerovo Regional Clinical Hospital', Kemerovo, Siberia
  - RSBIH 'Belgorod Regional Clinical Hospital of Saint Ioasaf', Belgorod
  - SBHI, Moscow
  - SBIH of Moscow region "Moscow Regional Scientific & Research, Moscow
  - SBEI HPE 'Rostov State Medical University' of the MoH of the RF, Rostov-on-Don
  - State Budgetary Institution of Healthcare of Yaroslavl region 'Clinical Hospital # 2', Yaroslavl
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Jeddah, Mecca Region
  - King Saud University, Riyadh
- Serbia (3):
  - Clinic of Neurology and Psychiatry for Children and Youth, Belgrade, Balkans
  - University Children Hospital, Belgrade, Balkans
  - Mother and Child Health Care Institute of Serbia ,,Dr Vukan Cupic'', Belgrade, Balkans
- Narodny ustav detskych chorob, Bratislava, Slovakia
- Spain (4):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
- Tunisia (3):
  - Hopital Razi, Manouba, Mannouba
  - Hôpital Fattouma Bourghiba, Monastir
  - Hôpital Habib Bourguiba, Sfax
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty Clinical Research Unit, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Izmir Dr. Behcet Uz Cocuk Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/